CLINICAL TRIAL: NCT03568968
Title: A Randomized Controlled Trial of Nicotinamide Riboside Supplementation in Early Parkinson's Disease: the NOPARK Study
Brief Title: A Randomized Controlled Trial of Nicotinamide Riboside Supplementation in Early Parkinson's Disease
Acronym: NOPARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other); Ostfold Hospital Trust (Other); Førde Hospital Trust (Other); Helse Fonna (Other); Molde Hospital (Other); Bodø sykehus (Unknown); Sorlandet Hospital HF (Other Government); Drammen sykehus (Other); University Hospital of Northern Norway, Tromsø, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/2083
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; NAD metabolism; Mitochondria; Nicotinamide Riboside
MeSH Terms: conditions — Parkinson Disease | interventions — nicotinamide-beta-riboside; NAD

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded study. N = 400 participants are randomized in a 1:1 ratio to either nicotinamide riboside (500 mg x 2 per day) or placebo.
Who Masked: Participant, Investigator
Masking Description: Study participants and investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (Experimental): nicotinamide riboside, 1000mg daily for the duration of the trial (52 weeks). Dosage form is capsules.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo Comparator (Placebo Comparator): Placebo capsules, no active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside 500mg administered two times a day. Given as capsules. Duration of the trial; 52 weeks.
  Other Names: NR, NAD, TruNiagen
  Arms: Nicotinamide Riboside
Other: Placebo — Placebo drug, administered two times a day. Given as capsules. Duration of the trial; 52 weeks.
  Arms: Placebo Comparator

SUMMARY:
NOPARK is a double-blinded randomized controlled phase II trial, with the aim to assess the efficacy of nicotinamide adenine dinucleotide (NAD)-replenishment therapy in the form of oral nicotinamide riboside (NR) in delaying the progression of early Parkinson's disease (PD). A total of 400 persons with early stage Parkinson's disease will be enrolled, randomized on nicotinamide riboside (NR) 500mg x 2 per day or placebo, and followed for 52 weeks.

DETAILED DESCRIPTION:
NOPARK is a multi-center, double-blinded randomized controlled trial, with the aim to assess the efficacy of NAD-replenishment therapy in the form of oral nicotinamide riboside (NR) in delaying the progression of early Parkinson's disease (PD). Individuals with PD (n = 400) will be recruited from multiple centers across Norway. Eligible participants must have been diagnosed with PD within 2 years of study enrollment and meet the trial's inclusion criteria. All participants will be given a standard PD-treatment regimen comprising selegiline 10 mg/day and oral levodopa (Sinemet or Madopar) at a dose of 100mg x 3, 150mg x3, or 200mg x 3 per day. The PD-treatment regimen will be frozen at baseline and remain stable throughout the duration of the study. At baseline, participants will be randomized on a 1:1 ratio on either nicotinamide riboside (NR) 500mg x 2 per day or placebo. Both the participants and the investigators will be blinded. The trial duration will be 52 weeks, during which participants will be assessed at baseline, 13, 26, 39 and 52 weeks. Measures include clinical evaluation using established scales for motor and non-motor dysfunction, as well as quality of life, 123I-N-ω-fluoropropyl-2β-carbomethoxy-3β-(4-iodophenyl) nortropane ([¹²³I]FP-CIT) single photon emission tomography (DaTscan), magnetic resonance imaging (MRI) of the brain, blood safety tests, and blood sampling for metabolomics, transcriptomics, and other exploratory analyses. The primary outcome of the study is the total score of the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of idiopathic PD according to the MDS clinical diagnostic criteria for Parkinson's disease
* [¹²³I]FP-CIT single photon emission CT (DaTscan) confirming nigrostriatal degeneration
* Diagnosed with PD within 2 years from enrolment
* Hoehn and Yahr score < 3 at enrolment
* Optimal symptomatic therapy, not requiring adjustments, for at least 1 month.
* Age equal to or greater than 35 years at time of enrolment.

Exclusion Criteria:

* Dementia or other neurodegenerative disorder at baseline visit
* Diagnosed with atypical parkinsonism or vascular parkinsonism
* Any psychiatric disorder that would interfere with compliance in the study.
* Any severe somatic illness that would make the individual unable to comply and participate in the study.
* Use of high dose vitamin B3 supplementation within 30 days of enrolment
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
* Genetically confirmed mitochondrial disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Disease severity assessed by the total MDS-UPDRS (Movement Disorder Society Unified Parkinson's Disease rating Scale): sum of subsections I, II, and III | From baseline to the end of treatment at 52 weeks
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assesses motor and non-motor symptoms of PD through four parts, with individual items rated on a 0-4 scale. Subscores are summed to provide a total score ranging from 0 to 260, with higher scores indicating greater disability. The primary outcome will be the MDS-UPDRS Total Score (sum of parts I, II, and III).

SECONDARY OUTCOMES:
Severity of motor symptoms in PD. | From baseline to the end of treatment at 52 weeks
  Change from baseline in the MDS-UPDRS Part III in the ON-medication state.
Severity of dopaminergic nigrostriatal denervation, assessed by [¹²³I]FP-CIT single photon emission CT (DaTscan) | From baseline to the end of treatment at 52 weeks
  Change from baseline in the mean striatal binding ratio (SBR) of the putamen, bilaterally, as measured [¹²³I]FP-CIT Single-Photon Emission Computed Tomography (SPECT) Imaging of the Dopamine Transporter (DaT, DaTscan).
Severiy of non-motor symptoms in daily living in PD | From baseline to the end of treatment at 52 weeks
  Change from baseline in the MDS-UPDRS Part I in the ON-medication state
Severity of motor aspects of experiences of daily living in PD. | From baseline to the end of treatment at 52 weeks
  Change from baseline in the MDS-UPDRS Part II
Severity of non-motor symptoms of PD assessed by the Non-Motor Symptoms Assessment Scale | From baseline to the end of treatment at 52 weeks
  Change from baseline in the NMSS Score in the ON-medication state. Non-Motor Symptoms Scale (NMSS) has 30 items, score range is 0-360 with higher scores indicating a worse outcome.
Change in the clinical severity of cognitive decline assessed by the Montreal Cognitive Assessment (MoCA) scale | From baseline to the end of treatment at 52 weeks
  Montreal Cognitive Assessment (MoCA), score range is 0-30 with lower scores indicating a worse outcome.
Change in quality of life assessed by the EuroQuality of Life Five Dimensions (EQ-5D-5L) questionnaire. | From baseline to the end of treatment at 52 weeks
  Quality of Life assessment (EuroQuality of Life Five Dimensions - EQ-5D-5L).
Hoehn and Yahr stage of PD | From baseline to the end of treatment at 52 weeks
  Hoehn and Yahr scale distinguishes between five stages in PD: Stage 1: Unilateral disease; Stage 2: Bilateral disease without impairment of balance; Stage 3: Bilateral disease with postural instability but physically independent; Stage 4: Severe disability; still able to walk or stand unassisted; Stage 5: Confinement to bed or wheelchair unless aided.

OTHER OUTCOMES:
brain nicotinamide adenine dinucleotide (NAD) levels | From baseline to the end of treatment at 52 weeks
  Change from baseline in brain NAD/ATP-α ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex).
systemic nicotinamide adenine dinucleotide (NAD) metabolism | From baseline to the end of treatment at 52 weeks
  Change from baseline in the NAD metabolome in whole blood or PBMC, measured by liquid chromatography mass spectrometry (LC-MS): Nicotinamide adenine dinucleotide oxidized (NAD+), Nicotinamide adenine dinucleotide reduced (NADH), NAD+/NADH ratio, total NAD (sum of NAD+ and NADH), Nicotinamide adenine dinucleotide phosphate oxidized (NADP+), Nicotinamide adenine dinucleotide phosphate reduced (NADPH), NADP+/NADPH ratio, total NADP (sum of NADP+ and NADPH, 1-methyl nicotinamide (Me-Nam), nicotinic acid-adenine dinucleotide (NAAD), N1-methyl-2-pyridone-5-carboxamide (Me-2-PY), Nicotinamide (Nam), Nicotinamide N-oxide (Nam N-oxide), ADP-ribose (ADPR), Nicotinic acid riboside (NAR), Nicotinamide riboside (NR), Nicotinamide mononucleotide (NMN), Nicotinic acid (NA).
neurofilament light-chain (NfL) levels | From baseline to the end of treatment at 52 weeks
  Change from baseline in serum neurofilament light-chain (NfL) levels, measured by Simoa analysis.
Safety and tolerablity | From baseline to the end of treatment at 52 weeks
  Report of all Adverse Events (AE) of moderate or severe intensity and Serious Adverse Events (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (11):
- Norway (11):
  - Bodø Hospital, Bodø, Nordland
  - Arendal Hospital, Arendal
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital, Drammen
  - Førde sykehus, Førde
  - Haugesund Hospital, Haugesund
  - Molde sjukehus, Molde
  - Akershus university hospital, Oslo
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - Østfold Hospital, Fredrikstad, Østland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03568968/SAP_000.pdf